CLINICAL TRIAL: NCT05953506
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of HS-10506 in Healthy Subjects
Brief Title: Phase 1a Study in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10506-101
Record Dates: First submitted 2023-06-26; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: HS-10506, Phase 1, Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10506 (Experimental): Healthy participants will be enrolled in dose escalation cohorts. Healthy participants will be receive either HS-10506 or matching placebo on Day 1.
  Interventions: Drug: HS-10506
- HS-10506 Placebo (Experimental): Healthy participants will be enrolled in dose escalation cohorts. Healthy participants will be receive either HS-10506 or matching placebo on Day 1.
  Interventions: Drug: HS-10506 Placebo

INTERVENTIONS:
Drug: HS-10506 — HS-10506 will be administered orally once on Day 1.
  Arms: HS-10506
Drug: HS-10506 Placebo — Matching placebo will be administered orally once on Day 1.
  Arms: HS-10506 Placebo

SUMMARY:
A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Oral HS-10506 in Chinese Healthy Subjects.

DETAILED DESCRIPTION:
This is a phase 1a, first-in-human, double-blind, placebo-controlled clinical trial. The primary objective is to assess the safety, tolerability and pharmacokinetic of single dose HS-10506 in healthy subjects. The secondary objective is to observed pharmacokinetic parameters and metabolites after single dose of HS-10506.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged from 18 to 45 years
* Subjects need to fully understand the research content and process, as well as possible adverse reactions, and voluntarily signed Informed Consent Form
* Males' weight ≥ 50kg, females' weight ≥ 45kg, body mass index {BMI, BMI=weight/height 2 (kg/m2)} is controlled within the range of 18~28 (including the critical value)
* During the study and for 3 months after receiving the last dose of study drug, subjects must agree not to donate sperm or eggs, not to plan to have children, and to use an effective method of contraception

Exclusion Criteria:

* Has a history of chronic or serious disease from neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal muscle system, metabolic endocrine system, skin disease, blood system, immune system or tumor
* Has taken any drugs, including prescription drugs, over-the-counter drugs, herbal preparations, some health products or inhibitor/inducer of CYP3A4 or CYP3A5, within 2 weeks (or 5 half-lives) before screening and throughout the study period
* Has clinically significant ECG abnormalities, such as QT interval corrected according to Fridericia formula(QTcF), >450 ms (males), >470 ms (females)
* Has current manifestation of blood pressure or pulse abnormalities in resting state: such as systolic blood pressure <90 mmHg or ≥140 mmHg, diastolic blood pressure <60 mmHg or ≥90 mmHg, pulse <55 bpm or >100 bpm

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-07-17 (Estimated); Primary Completion 2023-12-24 (Estimated); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs), serious adverse events (SAEs) and adverse events leading to discontinuation from the study, and their correlation with the investigational drug | Screening until Trail phase (up to 5 weeks)
  The definition of adverse event [AE] is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The definition of serious adverse event [SAE] is any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.
Number of participants with clinically significant change from baseline in vital signs | From baseline to Day 3
Number of participants with clinically significant abnormalities in physical examination | From baseline to Day 3
Changes in 12-lead electrocardiogram from before to after dosing | From baseline to Day 3
  Descriptive statistics of heart rate, PR interval, QT interval, and QTcF for observed values and changes from baseline will be summarized at each scheduled time point.
Change in Stanford Sleepiness Scale score from before to after dosing | From baseline to 4 hours after dosing
  Stanford Sleepiness Scale（SSS） is a simple and accurate method used to assess sleepiness symptom. Respondents use the scale from 1 to 7 to indicate their current level of sleepiness. Higher scores mean a higher level of sleepiness. Descriptive statistics of SSS scores and changes from baseline will be summarized at each scheduled time point.

SECONDARY OUTCOMES:
Observed maximum plasma concentration (Cmax) | up to 48 hours after dosing
  Cmax will be obtained following administration of a single oral dose of HS-10506.
Time to reach maximum plasma concentration (Tmax) | up to 48 hours after dosing
  Tmax will be obtained following administration of a single oral dose of HS-10506.
Area under the concentration-time curve from time zero to last time of quantifiable concentration（AUC0-t） | up to 48 hours after dosing
  Area under the concentration-time curve from time zero to last time of quantifiable concentration（AUC0-t）will be obtained following administration of a single oral dose of HS-10506.
Area under the concentration-time curve from time zero to infinity（AUC0-∞） | up to 48 hours after dosing
  AUC0-t will be obtained following administration of a single oral dose of HS-10506.
Terminal Rate Constant（λz） | up to 48 hours after dosing
  Terminal Rate Constant（λz） will be obtained following administration of a single oral dose of HS-10506.
Elimination Halflife (T1/2) | up to 48 hours after dosing
  Elimination Halflife (T1/2) is the time measured for the concentration to decrease by one half，which will be obtained following administration of a single oral dose of HS-10506.
Apparent clearance（CL/F） | up to 48 hours after dosing
  CL/F will be obtained following administration of a single oral dose of HS-10506.
Apparent Volume of Distribution（Vd/F） | up to 48 hours after dosing
  Vd/F will be obtained following administration of a single oral dose of HS-10506.
  Time Frame: up to 48 hours after dosing
Mean Residence Time(MRT) | up to 48 hours after dosing
  RT will be obtained following administration of a single oral dose of HS-10506.